CLINICAL TRIAL: NCT02606825
Title: VILMA: Therapeutic Results in Acute Mieloblastic Leukemia in Patients Older Than 60 Years or Not Candidates for Intensive Chemotherapy
Brief Title: VILMA: Therapeutic Results in Acute Mieloblastic Leukemia in Patients Older Than 60 Years
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: VILMA
Record Dates: First submitted 2015-10-13; First posted 2015-11-17 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: AML

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry of AML patients > 60 years

SUMMARY:
This is a retrospective study to analyze the therapeutic results and clinical evolution all patients diagnosed with AML and aged ≥ 60años or not candidates for chemotherapy intensive, treated according to the different schemes available, including supportive care or palliative.

DETAILED DESCRIPTION:
Approximately in 6 months, collect and review the retrospective data.

During this period, and in order to ensure an excellent quality of the collected data, perform constant monitoring and real-time data received in 2 phases:

1. Monitoring "in situ" in the focal point: once the information is received before shall enter in the database, will be reviewed each case report data (CRD) for screening for inconsistencies and issue unresolved issues (queries) to sender data center. After entering the information in the database is carry out and resolve those queries that have arisen after consultation Data tables in order to locate inconsistencies or unavailable fields.
2. Telephone Monitoring: data shall be verified through telephone consultations all centers to verify and update recruitment and monitoring patients . To ensure the completion, accuracy and data quality is monitored by telephone at least 30% of registered patients.

   * Final statistical analysis (approximately 8 months from baseline).
   * Publication of results.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥60 years, diagnosed of AML or not candidates to intensive chemotherapy

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥60 years, diagnosed of AML or not candidates to intensive chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 3910 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Response Rate | 8 months
  The main objective of this study is to retrospectively evaluate the therapeutic results in the LMA in all patients older than 60 years or not candidates for intensive chemotherapy in different stages of the disease, regardless of the treatment received, and even if they do not have received (support or palliative treatment, exclusively

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital General Universitario de Alicante, Alicante
  - ICO-Hospital Germans Trias i Pujol, Badalona
  - Hospital General Universitari de Castelló, Castelló
  - Hospital San Pedro Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de Gran Canaria Doctor Negrín, Las Palmas
  - Hospital Lucus Augusti, Lugo
  - CIBERONC, Instituto Carlos III, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Univeristario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Complutense University, i+12, CNIO, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Instituto de Biomedicina, Seville
  - Hospital Clínico Universitario, INCLIVA Biomedical Research Institute, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

REFERENCES:
- [Derived] Martinez-Cuadron D, Serrano J, Gil C, Tormo M, Martinez-Sanchez P, Perez-Simon JA, Garcia-Boyero R, Rodriguez-Medina C, Lopez-Pavia M, Benavente C, Bergua J, Lavilla-Rubira E, Amigo ML, Herrera P, Alonso-Dominguez JM, Bernal T, Colorado M, Sayas MJ, Algarra L, Vidriales MB, Rodriguez-Macias G, Vives S, Perez-Encinas MM, Lopez A, Noriega V, Garcia-Fortes M, Ramos F, Rodriguez-Gutierrez JI, Costilla-Barriga L, Labrador J, Boluda B, Rodriguez-Veiga R, Martinez-Lopez J, Sanz MA, Montesinos P. Evolving treatment patterns and outcomes in older patients (>/=60 years) with AML: changing everything to change nothing? Leukemia. 2021 Jun;35(6):1571-1585. doi: 10.1038/s41375-020-01058-4. Epub 2020 Oct 19. PMID 33077867